CLINICAL TRIAL: NCT06985043
Title: The Effect of Vagus Nerve Stimulation on Lower Limb Muscle Strength and Balance in Nonelite Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Tuğçe Poyraz İşleyen, PT, Bahçeşehir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E-10840098-202.3.02-2218
Record Dates: First submitted 2025-04-15; First posted 2025-05-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Vagus Nerve Stimulations; Muscle Strength; Balance
Keywords: vagus nerve stimulations, nonelite athletes, muscle strength, balance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vagus nerve stimulation (Experimental): Auricular vagus nerve stimulation (AVNS) will be applied to both ears simultaneously, using a biphasic, asymmetric waveform with pulses of 300 microsecond duration and a frequency of 25 Hz, continuously for 20 minutes. The application will be performed in a single session and the follow-up time will be determined as 30 minutes.
  Interventions: Device: Auricular vagus nerve stimulation (AVNS)

INTERVENTIONS:
Device: Auricular vagus nerve stimulation (AVNS) — Auricular vagus nerve stimulation (AVNS) will be applied to both ears simultaneously, using a biphasic, asymmetric waveform with pulses of 300 microsecond duration and a frequency of 25 Hz, continuously for 20 minutes. The application will be performed in a single session and the follow-up time will be determined as 30 minutes.

SUMMARY:
Clinical Trials (Non-Randomized Controlled) The aim of this study is to evaluate whether vagus nerve stimulation can improve neuromuscular and functional outcomes in non-elite athletes aged 18-35 years living in Istanbul.

The main questions it aims to answer are:

Does vagus nerve stimulation improve neuromuscular performance? Does it have a positive effect on functional performance? Researchers will compare the vagus nerve stimulation group to a control group to see if the intervention leads to significant improvements in neuromuscular and functional outcomes.

Participants will: Be selected based on criteria including age (18-35 years), non-elite athletic status (minimum two months), exercising 2-5 days per week for approximately 3.2 hours on average Have a Body Mass Index (BMI) between 18.5-25 kg/m² Participate voluntarily Exclusion criteria include:Any disease affecting the inner or outer ear BMI below 18.5 kg/m² or above 25 kg/m²

DETAILED DESCRIPTION:
The vagus nerve (VN), the tenth cranial nerve, is a key component of the neuroendocrine-immune axis and plays a critical role in regulating autonomic functions such as cardiovascular, endocrine, respiratory, and digestive system activity through its extensive central and peripheral connections (1,2). Non-invasive vagus nerve stimulation (VNS), particularly through auricular stimulation, has been shown to modulate autonomic balance by reducing sympathetic activity, enhancing cardiac baroreflex sensitivity, and improving parasympathetic tone (3,4).

In the context of athletic performance, the autonomic nervous system's role in adaptation to training and recovery is well recognized (5). Post-exercise parasympathetic reactivation is increasingly used as a biomarker for recovery and performance enhancement. Auricular VNS (aVNS), by stimulating afferent auricular branches of the VN, may facilitate recovery by reducing exercise-induced fatigue, pain, and lactate accumulation, while improving parasympathetic activity (3). Importantly, these physiological effects have been observed without significant alterations in heart rate or blood pressure.

Balance training is a known contributor to improved functional performance in athletes, and neuromuscular control is essential for injury prevention and overall athletic capacity (6). Considering the limited research on the effects of aVNS on neuromuscular parameters such as muscle strength and balance response in non-elite athletic populations, this study aims to provide evidence on the efficacy of aVNS in this context.

This study is designed as a non-randomized controlled trial. Thirty non-elite athletes aged 18-35 years, who have been physically active for at least three months and currently exercise 2-5 days per week (averaging 3.2 hours per week), will be recruited. Eligible participants must have a BMI between 18.5 and 25 kg/m² and provide informed consent. Individuals with conditions affecting the inner or outer ear or BMI values outside the specified range will be excluded.

The intervention group will receive a single session of bilateral aVNS using a biphasic, asymmetric waveform at a frequency of 25 Hz, pulse width of 300 microseconds, applied continuously for 20 minutes. The post-intervention follow-up period will last 30 minutes (3).

Assessment Parameters

Demographic and Baseline Characteristics:

Collected via a structured interview, including age, gender, height, weight, weekly exercise volume, and auditory health status.

Balance Assessment:

Balance will be evaluated using the Biodex Balance System, which quantifies postural sway and center of pressure (COP) metrics. Tests will be performed under both eyes-open and eyes-closed conditions, with three trials conducted for each. Lower sway index values indicate better balance performance (7).

Muscle Strength Assessment:

Maximal isometric strength of the quadriceps femoris and hamstring muscles will be measured using a Hand-Held Dynamometer (HHD). For quadriceps testing, participants will be seated with knees flexed to 90°, and the dynamometer placed 1-2 cm above the malleoli. For hamstring assessment, participants will lie prone with knees flexed to 90°. The "make test" method will be used, where the participant applies maximal voluntary contraction against a stationary dynamometer held by the examiner. Each muscle group will be tested three times with 60-second rest intervals, and the average value will be used for analysis (8).

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18.5-25 kg/m²
* exercising for a total of 3 hours or more per week for at least three months

Exclusion Criteria:

* have a chronic musculoskeletal disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Muscle strenght | Baseline and after the vagus stimulation apply
  Muscle strength of quadriceps femoris and hamstring muscles will be evaluated by hand dynamometer.
Balance | Baseline and after the vagus stimulation apply
  Postural sway will be assessed by biodex balance with center of gravity characteristics anterior-posterior and lateral sway with eyes closed and open.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahcesehir university, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peller A, Garib R, Garbe E, Komforti D, Joffe C, Magras A, Trapuzzano A, Stock MS, Dawson NT. Validity and reliability of the NIH Toolbox(R) Standing Balance Test As compared to the Biodex Balance System SD. Physiother Theory Pract. 2023 Apr;39(4):827-833. doi: 10.1080/09593985.2022.2027584. Epub 2022 Jan 23. PMID 35068342
- [Background] Unver B, Bakirhan S, Karatosun V. Does a weight-training exercise programme given to patients four or more years after total knee arthroplasty improve mobility: A randomized controlled trial. Arch Gerontol Geriatr. 2016 May-Jun;64:45-50. doi: 10.1016/j.archger.2016.01.003. Epub 2016 Jan 6. PMID 26952376
- [Background] Hrysomallis C. Balance ability and athletic performance. Sports Med. 2011 Mar 1;41(3):221-32. doi: 10.2165/11538560-000000000-00000. PMID 21395364
- [Background] Hatik SH, Arslan M, Demirbilek O, Ozden AV. The effect of transcutaneous auricular vagus nerve stimulation on cycling ergometry and recovery in healthy young individuals. Brain Behav. 2023 Dec;13(12):e3332. doi: 10.1002/brb3.3332. Epub 2023 Nov 16. PMID 37974551
- [Background] Caliota A, Ozden AV, Ceylan I. Effects of a single session of noninvasive auricular vagus nerve stimulation on sports performance in elite athletes: an open-label randomized controlled trial. Expert Rev Med Devices. 2024 Mar;21(3):231-237. doi: 10.1080/17434440.2023.2299300. Epub 2023 Dec 30. PMID 38146234
- [Background] Yuan H, Silberstein SD. Vagus Nerve and Vagus Nerve Stimulation, a Comprehensive Review: Part I. Headache. 2016 Jan;56(1):71-8. doi: 10.1111/head.12647. Epub 2015 Sep 14. PMID 26364692
- [Background] Prescott SL, Liberles SD. Internal senses of the vagus nerve. Neuron. 2022 Feb 16;110(4):579-599. doi: 10.1016/j.neuron.2021.12.020. Epub 2022 Jan 19. PMID 35051375